CLINICAL TRIAL: NCT05808387
Title: The Effects of Resveratrol on Inhibitors of Apoptosis Proteins, on Soluble Receptors of Advanced Glycation End Products and on Sirtuins-1 and -3 in Postmenopausal Women With Coronary Artery Disease
Brief Title: The Effects of Resveratrol on Sirtuins and Apoptosis Biomarkers
Acronym: RE-AGES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, Associate Professor, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61901722.6.0000.0068
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease; Menopause; Endothelial Dysfunction
Keywords: Coronary artery disease; Menopause; Endothelial Dysfunction; Sirtuin; Receptors of advanced glycation end products; Apoptosis; Resveratrol; Polyphenols; Cardiovascular risk
MeSH Terms: conditions — Coronary Artery Disease | interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial, parallel and placebo-controlled.
Who Masked: Participant, Care Provider
Masking Description: Participants in the control group will receive capsules identical to those in the intervention group, but with cornstarch.
  The care provider and the participants do not have the information about which capsules the participant is taking, and do not have access to which groups the patients belong. Statistical analyses will be performed on a blinded database, i.e. without information of which groups the participants belong to.
  Only the principal investigator of the study has this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): Trans-resveratrol, 1000mg daily for 90 days.
  Interventions: Dietary Supplement: Resveratrol
- Control (Placebo Comparator): Starch, 1000mg daily for 90 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Trans-resveratrol, 1000 mg daily for 90 days
  Arms: Resveratrol
Dietary Supplement: Placebo — Starch, 1000 mg daily for 90 days
  Arms: Control

SUMMARY:
Cardiovascular diseases (CVD) and neoplasms are the main causes of death in Brazilian women. Coronary artery disease (CAD) and stroke were responsible for approximately 54% of deaths from CVD in this population. In Brazil, cancers were the second cause of death and in 2017 were responsible for 58% of deaths in women. CVD and cancer share some risk factors, and control of these factors is associated with a significant reduction in cancer incidence. These two causes of death, although apparently disparate, share similar lifestyles and health risk factors, suggesting some common pathways and basic molecular networks. In women, the presence of estrogen has protective effects against atherosclerosis and, with the decline in hormone production at menopause, the incidence and prevalence of CAD increase substantially. Although the estrogen pathway is supposed to have a central effect on this increased risk, it is still debated whether other non-estrogenic mechanisms are related, since hormone replacement alone does not reduce cardiovascular events. Sirtuins and soluble advanced glycation product receptors (sRAGE) are associated with increased vascular protection, while the role of apoptosis inhibiting proteins, a pathway linked to increased cancer incidence, is still unclear in the context of atherosclerosis. Resveratrol is a key activator of sirtuins and potentially modulates these metabolic pathways, reducing cardiovascular risk. This randomized, double-blind, parallel, placebo-controlled clinical trial will be carried out in 80 postmenopausal women with CAD to analyze the effect of treatment with resveratrol on serum concentration and gene expression of sirtuins-1 -3, in the serum sRAGE concentration and in the gene expression of apoptosis inhibitory proteins.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the influence of sirtuins stimulation by resveratrol on inhibitors of apoptosis proteins gene expression of circulation angiogenic cells of postmenopausal women with stable coronary artery disease.

A randomized, double-blind, parallel, placebo-controlled clinical trial in postmenopausal women with CAD submitted to 90 days of daily resveratrol supplementation days of daily supplementation with 1000 mg of resveratrol. Eighty women aged ≥55 years, with overweight or obesity grade 1 (BMI between 25 and 35 kg/m2) will be selected. The participants will be randomized into two groups, control (CON) and resveratrol (RES). After the screening, the participants will undergo the first clinical and laboratory evaluation including lipid and glucose metabolism, inflammatory biomarkers, serum concentrations and gene expression of sirtuin-1 and sirtuin-3 and soluble receptor of advanced glycation end products, and the gene expression of inhibitors of apoptosis proteins.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women;
* Diagnosed coronary artery disease;
* Stable coronary disease;

Exclusion Criteria:

* hypo or hyperthyroidism,
* rheumatic disease,
* use of alcohol,
* hepatic failure,
* renal failure
* hormone replacement therapy
* use of insulin

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Sirtuin-1 and sirtuin-3 | 90 days
  Serum concentrations and gene expression
Inhibitors of apoptosis proteins | 90 days
  Gene expression of Bcl-2, XIAP, c-IAP1, and survivin
sRAGE | 90 days
  Serum concentrations and gene expression

SECONDARY OUTCOMES:
Inflammation | 90 days
  Serum concentrations of proinflammatory cytokines
Cardiometabolic risk factors | 90 days
  Lipid and glucometabolic profiles
Anthropometric measures | 90 days
  BMI, skinfold thickness, and body composition

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Mansur, PhD, Principal Investigator — InCor Heart Institute
Locations (1):
- INCOR- Heart Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No